CLINICAL TRIAL: NCT03764605
Title: Metformin vs Tolvaptan for Treatment of Autosomal Dominant Polycystic Kidney Disease. A Phase 3a, Indipendent, Multicentre, Two Parallel Arms, Randomized Controlled Trial
Brief Title: Metformin vs Tolvaptan for Treatment of Autosomal Dominant Polycystic Kidney Disease
Acronym: METROPOLIS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Loreto GESUALDO, Head of Nephrology, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudract2018-000477-77
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Metformin; Tolvaptan

STUDY DESIGN:
Intervention Model Description: Trial will enroll 150 subjects affected by Type I-truncating ADPKD. Their eligibility will be confirmed by the mean of eGFR calculated from the 2 pre-treatment serum creatinine assessments. Once eligibility is assessed, patients will undergo kidneys CTscan. Randomization visit will occur on Day -29. During this visit patients will be randomized (1:1) to each arm of treatment and will start IMP titration. Subjects not tolerating the minimum IMP dose will be considered "Titration failures" and will complete End of Treatment (EoTx) visit and will be followed up after 7 days by phone call. Subjects tolerating the minimum IMP dose enter the unblind run-in period during which, subjects will continue on a stable IMP dose to confirm tolerability over a longer period. At the end of the run-in period subjects not tolerating the minimum IMP dose will be considered "Run-in failures" and will complete EoTx visit. Subjects completing the run-in will start the open-label 24 months treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Patients will take metformin starting from 500 mg a day. They will up-titrate every week, if tolerating IMP, adding one 500 mg dose 8 hours after the former, till reaching 500 mg thrice a day.
  The minimum tolerated dose requested in order to be admitted to the study is 500 mg twice a day.
  Those reaching eGFR<45 ml/min will reduce the dose by one third. Those reaching eGFR<30 will drop out the study.
  Interventions: Drug: Metformin
- Tolvaptan (Active Comparator): Patient will start Tolvaptan in a split dose regimen 45 mg as first dose, followed by 15 mg 8 hours later. Those tolerating this dose will uptitrate to 60/30 mg and then to 90/30 mg a day. Those not tolerating 45/15 mg a day will drop out.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Metformin — Patieny will be treated by using Metformin from 500 mg a day to 500 mg thrice a day.
  Other Names: Zuglimet
  Arms: Metformin
Drug: Tolvaptan — Patients will be treated with tolvaptan from 45 mg + 15 mg a day to 90 mg + 30 mg a day
  Other Names: Jinarc
  Arms: Tolvaptan

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common inherited renal disorder occurring in 1:400-1:1.000 live births and affects 4 to 6 million persons worldwide and about 205.000 people in Europe (EU). This figure is equivalent to 4 in 10.000 people and thus below the prevalence threshold of 5 in 10.000 used to designate a disease as rare in EU.

Renal cyst development and expansion in ADPKD involves both fluid secretion and abnormal proliferation of cyst-lining epithelial cells. The chloride channel of the cystic fibrosis transmembrane conductance regulator (CFTR) participates in secretion of cyst fluid, and the mammalian target of rapamycin (mTOR) pathway may drive proliferation of cyst epithelial cells. CFTR and mTOR are both negatively regulated by AMP-activated protein kinase (AMPK). Metformin, a drug widely used, is a pharmacological activator of AMPK. The investigators found that metformin stimulates AMPK, resulting in inhibition of both CFTR and the mTOR pathways. Metformin induces significant arrest of cystic growth in both in vitro and ex vivo models of renal cystogenesis. In addition, metformin administration produces a significant decrease in the cystic index in two mouse models of ADPKD. These results suggest a possible role for AMPK activation in slowing renal cystogenesis as well as the potential for therapeutic application of metformin in the context of ADPKD.

Thus this study aims to evaluate metformin efficacy in slowing renal cystogenesis in ADPKD as compared to the actual gold standard (Tolvaptan).

DETAILED DESCRIPTION:
Objective of the study is to assess if a two-year course of 1500 mg oral metformin is effective and safe in treatment of ADPKD, as compared to the actual gold-standard therapy, tolvaptan (Jinarc®) This is a phase 3a, independent, multi-centre, parallel arms, randomized controlled trial comparing efficacy and safety of metformin and tolvaptan in ADPKD.

This trial will enroll approximately 150 tolvaptan and metformin naïve subjects affected by Type I-truncating ADPKD, as these subjects have grater probability of progression.

The trial contemplates a 2 weeks screening period (included in a 9 months total recruitment period) during which 3 visits have to be collected (the 1st and the 2nd in three days, and the 3rd after biochemical analyses performed during the first two visits have been reviewed). The subject's eligibility for the trial will be confirmed by the mean of eGFR calculated from the 2 pre-treatment, central-lab, serum creatinine assessments. Longer screening periods (up to 4 additional weeks) are acceptable for subjects needing stabilization after changing or discontinuing other treatments, especially anti-hypertensives and diuretics.

Once eligibility is assessed, patients will undergo non-contrast enhanced CT-scan of kidneys (if not performed within six months prior to randomization).

Randomization visit will occur on Day -29. During this visit patients will be randomized (in a ratio 1:1 tolvaptan:metformin) to each arm of treatment and will start an IMP titration period (3 weeks from -28 to -8). Subjects not tolerating the minimum IMP dose will be considered "Titration failures" and will complete End of Treatment (EoTx) visit assessments and will be followed up after 7 days by phone call to assess any ongoing AEs. Subjects tolerating the minimum IMP dose enter the unblind run-in period (1 week from Day -7 to -1). During the "Run-in" phase, subjects will continue on a stable IMP dose to confirm tolerability over a longer period. At the end of the run-in period (Day -1), subjects not tolerating the minimum IMP dose will be considered "Run-in failures" and will complete EoTx visit assessments and will be followed up after 7 days by phone call to assess any ongoing AEs. Subjects completing the run-in will start the open-label 24 months treatment period, during which visits will be collected three-monthly. At the end of the 24th month, and in case of early treatment cessation, follow-up period (3 weeks from +8 to +21) will start, during which 2 visits have to be collected. No IMP will be administered during this period.

This trial will enroll approximately 150 tolvaptan and metformin naïve subjects and will be conducted in about 11 Italian Hospital Nephrology Departments The investigators plan to recruit a total of 150 patients which are currently within the reach of the network coordinated by the proponent and composed by 11 Nephrology Centres. This network treats a total of 1500 (already genetically studied) patients of which the investigators expect (based on standard response rates recognized in the population) acceptance to participate in the study to a value of approximately 40% of patients that will be then allocated to the experimental and control intervention.

The selected sample is adequate to evaluate a significant reduction in the slope of eGFR at 2 years by 10%, which is a clinically relevant piece of information at the current state of knowledge, as well as a complete assessment of the benefits-harms trade-off of the two interventions.

The trial has a 36 months overall duration, that include a 9 months recruitment period; has a 2 weeks duration, it is included in the 9 months recruitment period. The treatment period has a 25 months duration. Each month lasts 28 days. It includes the 3 weeks titration period and the 1 week run-in period.

The post-treatment follow-up: lasts 21 days. The total Study Duration is of about 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 50 years
2. eGFR (CKD-EPI) ≥ 45 ml/min/1,73 m2
3. Genetic Diagnosis of Type I ADPKD truncating mutation
4. Signed and dated informed consent

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of IMP. If employing birth control, 2 of the following precautions must be used: vasectomy of partner, tubal ligation, vaginal diaphragm, intrauterine device, birth control implant, condom, or sponge with spermicide. Non-childbearing potential in women is defined as female subjects who are surgically sterile (ie, have undergone bilateral oophorectomy or hysterectomy) or female subjects who have been postmenopausal for at least 12 consecutive months.
2. Women who are breast-feeding and/or who have a positive pregnancy test result prior to receiving investigational medical product (IMP).
3. Treatment with acarbose, guar gum, cimetidin, phenprocoumon, oral anticoagulants, thrombolytic drugs, diuretics, ranolazin, cephalexin.
4. Evidence of active systemic or localized major infection at the time of screening.
5. Hepatic impairment or liver function abnormalities other than that expected for ADPKD with typical cystic liver disease during the screening period as defined by:

   * AST O ALT >8x UNL
   * AST O ALT >5x UNL >2 WEEKS
   * AST O ALT >3x UNL E BT >2x UNL OR INR >1,5
   * AST O ALT >3x UNL E SIGNS AND SYMPTOMS OF LIVER DAMAGE (fatigue, anorexy, nausea, vomiting, right hypocondrium pain, fever, jaundice, skin rash, itching)
6. Acute or chronic disease causing tissue hypoxia (e.g.: myocardial failure, severe arythmias, myocardial infarction, respiratory failure, liver failure, alcohol acute intoxication, alcoholism, dehydration).
7. Previously diagnosed diabetes already in treatment with other hypoglycemic drugs.
8. Ongoing breast feeding.
9. Use of any other investigational drug or treatment up to 4 weeks before enrollment and during the treatment phase.
10. Known hypersensitivity to metformin and its derivatives.
11. Psychiatric disorders and any condition that might prevent full comprehension of the purposes and risks of the study.
12. Malignancies within three years before enrolment in the study.
13. HIV, HBV, HCV infection.
14. Urinary tract obstruction.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (estimated by CKD-Epi formula) variation | 25 months
  Primary outcome of the study is to evaluate the difference between Metformin and Tolvaptan in annualized slope of eGFR (CKD-EPI) for individual subjects, that will be calculated using an appropriate baseline and post-randomization assessment.

SECONDARY OUTCOMES:
Total Kidney Volume variation (measured by non contrast enhanced Kidney CT scan) | 25 months
  The key secondary endpoint is the percent change from baseline in htTKV as measured by CT-scan at 24 months.

OTHER OUTCOMES:
Blood pressure | 36 months
  mmHg
Post void body weight | 36 months
  Kg
Change from serum creatinine baseline | 36 months
  mg/dl
Serum sodium | 36 months
  mg/dl
Blood venous gas lactate levels | 36 months
  mmol/l
Bolood Glucose levels | 36 months
  mg/dl
Vitamin B12 deficency | 36 months
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, Principal Investigator — AOUConsorziale Policlinico di Bari
Locations (2):
- Italy (2):
  - AOUC "Policlinico", Bari
  - AOUConsorziale Policlinico Di Bari, Bari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT03764605/Prot_SAP_000.pdf